CLINICAL TRIAL: NCT01253018
Title: Evaluation of Robot Assisted Neuro-rehabilitation
Acronym: SRT3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Massachusetts Institute of Technology (Other); University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6935-R
Record Dates: First submitted 2010-11-24; First posted 2010-12-03 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: stroke; robotics; upper extremity rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot Therapy (Experimental): 12 weeks of robotic therapy
  Interventions: Behavioral: Robot Therapy
- Transition to Task Training (Active Comparator): 12 weeks of task specific practice combined with robotic therapy
  Interventions: Behavioral: Transition to Task Training

INTERVENTIONS:
Behavioral: Robot Therapy — Robot assisted arm exercise for 60 minutes progressing each month through three robot modules: wrist, planar, and alternating sessions on the wrist and planar robot 3x/week for 12 weeks.
  Other Names: Upper extremity (UE) robot-assisted exercise
  Arms: Robot Therapy
Behavioral: Transition to Task Training — Robot therapy as described for 45 minutes and 15 minutes of task specific arm exercise using the hemiparetic arm 3x/week for 12 weeks.
  Arms: Transition to Task Training

SUMMARY:
Robotic devices are capable of providing therapy to the arm of patients with weakness due to stroke. Robotic therapy improves some aspects of stroke related arm weakness, but the use of the weak arm for real life situations often remains limited. The goal of this study is to determine the best way to use robotic devices and functional task training to improve the use of the stroke affected arm for real life situations. A secondary goal of this study is to determine how or if specific areas of the brain are excited before and after training. The use of a safe and painless magnetic field directed at the brain called transcranial magnetic stimulation (TMS) will be used at set intervals to gain a better understanding of brain activity during recovery.

DETAILED DESCRIPTION:
After obtaining informed consent, participants will undergo 3 sessions of baseline testing using upper extremity motor assessments of the shoulder, elbow, wrist, thumb and grip. Upper extremity kinematic and strength testing will be performed with the rehabilitation robots in measurement mode. The rehabilitation robot modules include the wrist, the planar (shoulder-elbow), and alternating wrist and shoulder-elbow robot. These robotic devices are cleared for marketing as a registered medical device under U.S. FDA regulations and are listed with the FDA both as an evaluation devices and as therapy devices.

Patients will be randomized to receive 12 weeks of robotic therapy sessions or 12 weeks of robot therapy combined with transition to task therapy. Study interventions will occur 3 times a week for 12 weeks. Robot therapy will consist of a progression through three robot modules: wrist, planar, and alternating wrist and shoulder-elbow robot. The progression will be sequential with four weeks of training on each robotic device. All participants will complete a motor activity log during this intervention phase.

TMS is being used for physiological measurement and evaluations will be conducted with each participant at baseline, week one, week five, eight, and final. TMS will also occur during the follow-up on week twenty-four.

Disability and depression questionnaires, upper extremity measures and evaluations of functional performance will be conducted during the study at baseline, and at training completion (visit 36). Patients will return twelve weeks after the end of the training period to determine whether any observed improvements persist.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined, unilateral, hemiparetic stroke with radiologic exclusion of other possible diagnoses
* Adequate language, and cognitive function to participate in training, testing, and informed consent process
* The study arm of the participant will present with moderate to severe dysfunction based on Fugl-Meyer Motor Assessment range of 7 to 38
* Stroke onset greater than 6 months for ischemic stroke and greater than 1 year for hemorrhagic stroke
* Men or women over 21 years of age

Exclusion Criteria:

* Seizures or treatment with anticonvulsant medications within the last 10 years (This criteria does not preclude participation in the study, but does preclude participation in the TMS testing)
* Treatment with any medications known to interfere with brain stimulation: any medication with central nervous system depressant activity, including, but not limited to benzodiazepines, barbiturates, and neuroleptics (This criteria does not preclude participation in the study, but does preclude participation in the TMS testing)
* Serious complicating medical conditions, contractures or orthopedic problems in the study arm limiting the range of joint movement for the study positions
* Visual loss such that the participant cannot see the test patterns on the monitor of the training robot computer
* Botox injection to the study arm within 3 months of enrollment or during the study period
* Any change in the exercise regime involving the study arm. This includes starting any new exercise or discontinuing any current exercise regimen

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2015-01-16 (Actual); Study Completion 2015-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T. Bever, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

REFERENCES:
- [Result] Conroy SS, Wittenberg GF, Krebs HI, Zhan M, Bever CT, Whitall J. Robot-Assisted Arm Training in Chronic Stroke: Addition of Transition-to-Task Practice. Neurorehabil Neural Repair. 2019 Sep;33(9):751-761. doi: 10.1177/1545968319862558. Epub 2019 Jul 22. PMID 31328671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2011 and March 2014. The study location was a clinical research setting within the Veterans Affairs Maryland Health Care System.
Pre-assignment Details: 14 enrolled participants were withdrawn prior to randomization due to not meeting FM inclusion criteria, or due to medical or social issues.
Groups:
- Robot Therapy: 12 weeks of robot-assisted upper extremity exercise using 2 different robots in a sequential 4 week progression in 3 distinct modules: wrist, shoulder-elbow and alternating sessions of wrist and shoulder-elbow robot. Sessions were 3x/week x 60 minutes.
- Transition to Task Training: 12 weeks of robot-assisted upper extremity exercise as described in robot therapy group combined with transition to task (TTT) practice using the hemiparetic arm for functional activities. Session were 3x/week x 60 minutes (45 minutes robot therapy + 15 minutes TTT)
Period: Overall Study
Arm/Group | Robot Therapy | Transition to Task Training
Started | 22 | 23
Completed | 18 | 21
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Robot Repair Issues | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Age, gender, race/ethnicity, type of stroke.
Groups:
- Robot Therapy: 12 weeks of robot-assisted upper extremity exercise using three upper extremity robot modules: wrist, planar, and alternating wrist and planar robot each in a 4 week sequential progression. Sessions 3x/week x 60 minutes
- Transition to Task Training: 12 weeks of robot-assisted upper extremity exercise as described in Robot Therapy combined with transition to task (TTT) practice of functional activities using the hemiparetic arm. Sessions were 3x/week x 60 minutes (45 min robot therapy + 15 min TTT)
- Total: Total of all reporting groups
Arm/Group | Robot Therapy | Transition to Task Training | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.2) | 56.4 (12.7) | 56.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 14 | 21
  Black or African American | 14 | 8 | 22
  Asian Indian | 0 | 1 | 1
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45
Type of Stroke [Number; unit: participants]
  Ishemic | 18 | 19 | 37
  Hemorrhagic | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Motor Upper Extremity Assessment
Description: This is a stroke-specific measure of impairment of the upper extremity that has been shown to be valid and reliable with high inter-rater and test-retest reliability. It provides a direct-observational assessment of volitional movement and motor impairment related to reflexes, sensation, and abnormal synergies. Each item on the FM is rated on a three-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully). The scale ranges from 0-66 with higher scores representing less motor impairment.
Time Frame: Baseline, 12 week, and 24 week retention
Population: All participants completing the 12 week intervention including evaluations at baseline, weeks 4, 8, 12 and at the 24 week retention evaluation. 1 participant in each group did not return for retention and were not included in the retention analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot Therapy | Transition to Task Training
Number analyzed (Participants) | 19 | 22
units on a scale
  Change BL to 12 weeks | 2.7 (3.0) | 3.7 (3.4)
  Change BL to 24 weeks | 3.7 (4.6) | 3.5 (4.0)
Statistical Analysis 1: Comparison: Robot Therapy vs Transition to Task Training; Sample size and power calculations were performed based on the difference in the FM score between the two groups with an assumed within group SD of 15.9, the correlation of 0.5 among repeated measures. 30 subjects enrolled in each arm of the study would give 80% power for detecting a difference of 8 points on the FM. Two sample t-tests were conducted to compare changes in FM between the two interventions groups at final training (12 week); Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Robot Therapy vs Transition to Task Training; Two sample t-tests were conducted to compare changes in FM between the two interventions groups at retention (24 weeks); Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Motor Cortex Excitability Via Transcranial Magnetic Stimulation (TMS)
Time Frame: week 12
Population: The severity of the patients enrolled in the study were such that TMS did not evoke the number of motor action potentials needed for analysis.
Arm/Group | Robot Therapy | Transition to Task Training
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: The Wolf Motor Function Test (WMFT) examines UE function based on task performance time, quality of movement, and ability to hold a weight. Functional use and speed of movement are based on fifteen timed activities and two strength activities. It has high inter-rater reliability, internal consistency, and test-retest reliability. Timed tasks that cannot be completed default to a time score of 120 seconds. Faster times or a lower score in seconds represent better function. Improvement is represented by a decreased time to complete the tasks therefore a negative change score from baseline to follow-up indicates improvement.
Time Frame: Baseline, 12 week, and 24 week retention
Population: All participants completing the 12 week intervention including evaluations at baseline, weeks 4, 8, 12 and at the 24 week retention evaluation. The change score from baseline to the final (12 week) evaluation was examined. 1 participant in each group did not return for retention and were not included in the retention analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robot Therapy | Transition to Task Training
Number analyzed (Participants) | 19 | 22
seconds
  Change BL to 12 weeks | -5.1 (6.2) | -9.4 (10.3)
  Change BL to 24 weeks | -7.6 (9.8) | -8.6 (11.8)
Statistical Analysis 1: Comparison: Robot Therapy vs Transition to Task Training; Two sample t-tests were conducted to compare changes in WMFT between the two interventions groups at final training 12 week; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Robot Therapy vs Transition to Task Training; Two sample t-tests were conducted to compare changes in WMFT between the two interventions groups at retention 24 weeks; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Stroke Impact Scale: Hand Subscale
Description: The Stroke Impact Scale (SIS) is a self-report structured interview consisting of eight domains designed to assess changes in impairment, disabilities, and handicap following stroke that contribute to quality of life. It has been tested and found to be reliable, valid, and sensitive to change in the stroke population. There are four physical domains that that can be analyzed separately. The hand domain was analyzed for this study and the scores for this domain range from 0-100. Higher scores indicate greater function.
Time Frame: Baseline, 12 week and 24 week retention
Population: All participants completing the 12 week intervention including evaluations at baseline, weeks 12 and the 24 week retention evaluation. The change score from baseline to the final (12 week) evaluation was examined. 1 participant in each group did not return for retention and were not included in the retention analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot Therapy | Transition to Task Training
Number analyzed (Participants) | 19 | 22
units on a scale
  Change BL to 12 weeks | 5.8 (14.3) | 15.5 (20.4)
  Change BL to 24 weeks | 7.8 (12.0) | 13.8 (16.5)
Statistical Analysis 1: Comparison: Robot Therapy vs Transition to Task Training; Two sample t-tests were conducted to compare changes in SIS Hand between the two interventions groups at final training week 12; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Robot Therapy vs Transition to Task Training; Two sample t-tests were conducted to compare changes in SIS Hand between the two interventions groups at retention week 24; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8.5 months
Arm/Group | Robot Therapy | Transition to Task Training
Serious Adverse Events (participants affected / at risk) | 3/21 | 4/22
Other Adverse Events (participants affected / at risk) | 0/21 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robot Therapy (N=21) | Transition to Task Training (N=22)
Stent Placement (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fib (Cardiac disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Hospitalization to r/o new CVA (Nervous system disorders) | 0 (0) | 2 (2) — Hospital findings negative for new CVA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robot Therapy (N=21) | Transition to Task Training (N=22)
Fall at home with resulting fx to study arm (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)

LIMITATIONS AND CAVEATS:
The amount of change on our primary outcome measure (FM) for this population of stroke survivors with moderated to severe upper extremity motor impairment was less than predicted (4 points vs. 8) resulting in the study groups being underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes